CLINICAL TRIAL: NCT06482788
Title: Perioperative Treatment of Resectable Adenocarcinoma of Esophagogastric Junction by Immunotherapy (Adebrelimab) Combined With Chemotherapy (XELOX): a Prospective, Single-center, Feasibility Study
Acronym: AEGIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTS-023
Record Dates: First submitted 2024-05-22; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-05

CONDITIONS: Esophagogastric Junction Adenocarcinoma
MeSH Terms: interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): Patients will receive Immunotherapy (Adebrelimab, PD-L1 inhibitor) combined with XELOX chemotherapy (Capecitabine + Oxaliplatin) therapy in four 3-week treatment cycles with imaging assessment every 2 cycles. After treatment response evaluation, patients will receive resection within 4-8 weeks. Following surgery, patients will receive four further 3-week cycles of Adebrelimab + XELOX after 4-12 weeks of resection. Patients will then receive 10 additional 3-week treatment cycles with Adebrelimab alone.
  Interventions: Drug: Adebrelimab (anti-PD-L1) + XELOX

INTERVENTIONS:
Drug: Adebrelimab (anti-PD-L1) + XELOX — Adebrelimab: 1200mg, i.v., each infusion lasts 30-60 minutes and is administered on the first day of each cycle (3 weeks).
  Capecitabine: 1000mg/m2 , bid, orally, from day 1 to day 14 of each cycle (3 weeks).
  Oxaliplatin: 130mg/m2, i.v., each infusion is administered on the first day of each cycle (3 weeks).

SUMMARY:
The purpose of this study is to explore the effectiveness and safety of immunotherapy (Adebrelimab, a PD-L1 inhibitor) combined with standard chemotherapy (XELOX) in the perioperative treatment of resectable esophagogastric junction adenocarcinoma.

DETAILED DESCRIPTION:
The study will evaluate the efficacy and safety of the immunotherapy (Adebrelimab) combined with standard chemotherapy (XELOX) in the perioperative treatment of resectable esophagogastric junction adenocarcinoma. Potential study participants will be assessed for eligibility during a 28-day screening period that includes central verification of clinical stage and eligibility. Eligible patients will be receive perioperative treatment with adebrelimab with XELOX. Location of the primary (GEJ type I vs. GEJ type II/III vs. stomach), and PD-L1-status (CPS≥5 vs. CPS<5). Microsatellite Instability (MSI-H vs MSI-L) will be will be given special attention.

ELIGIBILITY:
Inclusion Criteria:

* Sign on the informed consent form (ICF)
* Histologically confirmed esophagogastric junction Adenocarcinoma (AEG, Type Siewert I/II/ III), the stage is locally advanced cT1b-2N+ or T3-4Nany that the investigator judges it to be resectable (1. CT or MRI assessment shows no invasion of adjacent organs or tissues, 2. No peritoneal metastasis occurs, 3. There are surgical indications) (Note: If bone lesions are suspected, a bone scan is required; if peritoneal carcinomatosis is suspected, laparoscopy is required to confirm; if T3-T4 subjects have diffuse tissue types, diagnostic laparoscopy is also required))
* No previous systematic treatment
* At least one measurable lesion according to RECIST 1.1.
* ECOG PS: 0-1
* The functions of important organs meet the following requirements：Absolute neutrophil count ≥ 1.5 × 109/L； Platelet ≥ 100 × 109/L； Hemoglobin ≥ 90g / l; ALT and AST ≤ 2.5 times ULN; TBIL ≤ 1.5 times ULN; Serum creatinine ≤ 1.5 times ULN or creatinine clearance ≥ 60ml / min; INR ≤ 1.5, APTT ≤ 1.5 times ULN; No obvious abnormality on electrocardiogram.
* Male subjects and women of childbearing age must take contraceptive measures from the first dose to the last 3 months of use of the study drug.

Exclusion Criteria:

* Histologically confirmed Squamous cell carcinoma or mixed type.
* Distant metastasis: If peritoneal cancer or ascites is suspected by imaging, histological or cytological confirmation such as laparoscopic exploration is required.
* Medical history and complications: 1.Having contraindications to surgical resection of esophagogastric junction cancer 2.Having any known active autoimmune diseases 3.Having any complications that require systemic treatment with glucocorticoids such as prednisone (>10 mg/day) or have used immunosuppressive drugs within 14 days before the first dose
* Having received tumor vaccines or other immune-activating anti-tumor drugs (such as interferon, interleukin, thymosin or immune cell therapy) within 1 month before the first dose 4.Having participated in other clinical trials or have received drug interventions from other clinical trials within 4 weeks before the first dose 5.Having other malignant tumors that need treatment 6.Having a history of severe cardiovascular disease 7.Having a known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
* Severe allergic reaction to drugs (Adbrelimab, Capecitabine, Oxaliplatin).
* The subjects were innate or acquired immunodeficiency (such as HIV), or active hepatitis (hepatitis B reference: HBsAg) positive; Hepatitis C reference: HCV antibody positive.
* According to the judgment of the researcher, the subject has other factors that may lead to the forced midway termination of this study, such as other serious diseases (including mental diseases) requiring combined treatment, serious laboratory abnormalities, accompanied by family or social factors, which will affect the safety of the subject, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (ITT) | From date of enrolment until surgical resection, an average of 3 months
  The proportion of subjects with no cancer cells in the primary tumor and lymph node specimens (ypT0N0)

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li Y, Cao Y, Wang X, Li C, Zhao L, Li H. Effects of perioperative treatment of resectable adenocarcinoma of esophagogastric junction by immunotherapy (Adebrelimab) combined with chemotherapy (XELOX): protocol for a single-center, open-labeled study (AEGIS trial, neoadjuvant immunochemotherapy). BMC Cancer. 2025 Feb 4;25(1):198. doi: 10.1186/s12885-025-13589-z. PMID 39905364